CLINICAL TRIAL: NCT03787160
Title: Determining the Effect of Probiotics on Microbiome and Volatile Organic Compounds in Patients After Surgical Repair of Congenital Diaphragmatic Hernia
Brief Title: Microbiome and Volatile Organic Compounds in Patients With CDH
Acronym: CDHVOCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: University of Rostock (Other)
Responsible Party: Principal Investigator, Warncke Gert, MD, Principal Investigator, Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 28-528 ex 15/16
Record Dates: First submitted 2018-07-10; First posted 2018-12-26 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: congenital diaphragmatic hernia; volatile organic compounds; microbiome; pulmonary function; multiple breath washout
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital | interventions — Functional Residual Capacity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDH Group (Active Comparator): 10 patients after surgical closure of CDH will undergo VOC profile analysis (2 breath samples) (initial VOC), fecal sampling for 16S rDNA based pyrosequencing (initial fecal microbiome) and deep induced sputum sampling for 16S rDNA pyrosequencing (initial pulmonary microbiome), bicycle spiroergometry to determine the maximum oxygen uptake (maximum oxygen uptake), body plethysmography, spirometry and N2-multiple breath washout testing to determine the functional residual capacity (functional residual capacity). Thereafter patients will receive probiotic treatment with OmniBiotic6 (R) (Allergosan, Graz, Austria) 1 sachet daily for 3 months (probiotic treatment). Three months after discontinuing probiotic treatment VOC testing (VOC probiotics), fecal microbiome sampling (fecal microbiome probiotics) and deep induced sputum testing (pulmonary microbiome probiotics) will be repeated and compared to the results of the initial tests.
  Interventions: Diagnostic Test: initial VOC; Diagnostic Test: initial fecal microbiome; Diagnostic Test: initial pulmonary microbiome; Diagnostic Test: Maximum oxygen uptake; Diagnostic Test: Functional residual capacity; Dietary Supplement: Probiotic treatment; Diagnostic Test: VOC probiotic; Diagnostic Test: Fecal microbiome probiotic; Diagnostic Test: Pulmonary microbiome probiotic
- Control Group (Other): 10 healthy controls (age and sex matched) will undergo VOC profile analysis (2 breath samples) (initial VOC), fecal sampling for 16S rDNA based pyrosequencing (initial fecal microbiome) and deep induced sputum sampling for 16S rDNA pyrosequencing (initial pulmonary microbiome), bicycle spiroergometry to determine the maximum oxygen uptake (maximum oxygen uptake), body plethysmography, spirometry and N2-multiple breath washout testing to determine the functional residual capacity (functional residual capacity).
  Interventions: Diagnostic Test: initial VOC; Diagnostic Test: initial fecal microbiome; Diagnostic Test: initial pulmonary microbiome; Diagnostic Test: Maximum oxygen uptake; Diagnostic Test: Functional residual capacity

INTERVENTIONS:
Diagnostic Test: initial VOC — Difference in VOC profile between patients with CDH and healthy controls (2 samples per patient will be obtained after obtaining informed consent).
Diagnostic Test: initial fecal microbiome — Difference of alpha and beta diversity and relative fecal bacterial abundance between patients with CDH and healthy controls (1 stool sample will be taken per patient after obtaining informed consent)
Diagnostic Test: initial pulmonary microbiome — Difference of alpha and beta diversity and relative pulmonary bacterial abundance between patients with CDH and healthy controls (1 deep induced sputum sample will be taken per patient after obtaining informed consent)
Diagnostic Test: Maximum oxygen uptake — Comparison of the maximum oxygen uptake (corrected for body weight and gender) as determined by bicycle spiroergometry between patients with CDH and healthy controls
Diagnostic Test: Functional residual capacity — FRC will be determined by spirometry, bodyplethysmography and N2-breath wash out method. FRC will be compared between patients after CDH and healthy controls.
Dietary Supplement: Probiotic treatment — CDH patients will receive OmniBiotic 6(R) (Allergosan, Graz, Austria) probiotic supplementation 1 sachet daily for 3 months.
  Arms: CDH Group
Diagnostic Test: VOC probiotic — Determination of the VOC profile 3 months after discontinuing probiotic treatment. Comparison to the profiles before the treatment.
  Arms: CDH Group
Diagnostic Test: Fecal microbiome probiotic — Determination of the fecal microbiome from 1 sample per patient (alpha and beta diversity, relative bacterial abundance at the genus level) 3 months after discontinuing probiotic treatment. Comparison to the profiles before the treatment.
  Arms: CDH Group
Diagnostic Test: Pulmonary microbiome probiotic — Determination of the fecal microbiome from 1 deep induced sputum sample per patient (alpha and beta diversity, relative bacterial abundance at the genus level) 3 months after discontinuing probiotic treatment. Comparison to the profiles before the treatment.
  Arms: CDH Group

SUMMARY:
Despite improved prenatal diagnostics and therapeutic possibilities, congenital diaphragmatic hernia (CDH) represents a cross-disciplinary challenge. With an incidence of 1:2000-1:5000, it is a common disease that effects centres of paediatrics and juvenile medicine. The etiology is still unclear. Patients with this diagnosis are usually affected by other comorbities such as failure to thrive, gastroesophageal reflux, funnel chest, etc. Depending on the extent of CDH, a more or less pronounced lung hypoplasia with functional impairment occurs. The health-relevant importance of the human microbiome is increasingly evident. While it was previously particularly associated with the gastrointestinal tract, other systems such as the pulmonary microbiome have become the focus of scientific interest.

Research into changes in the microbiome and volatile organic compounds (VOCs) could provide new insights into the underlying mechanisms and therapeutic measures of this disease.

DETAILED DESCRIPTION:
Aim: The aim of this study is to evaluate children who have been enrolled on the basis of a hernia, the pulmonary microbiome and the volatile organic compounds (VOCs) in the exhaled air and to compare them with a control group which does not have a chronic or acute lung disease. Furthermore, the lung function by spirometry, whole body plethysmography and "multiple breath washout" procedures be precisely recorded and a sports medical examination, including ergospirometry. In addition, any influence of probiotics on the pulmonary microbiome in children with diaphragmatic hernia will be investigated.

Study design: This is a prospective study in children who were treated surgically in early childhood for congenital diaphragmatic hernia. After an initial determination of the microbiome and the composition of volatile organic substances in breathing air and feces and a lung function measurement as well as sports medical examination, the study group receive a probiotic (Omnibiotics 6, obtained from the Allergosan Institute, food supplements) for 3 months. The microbiome and VOCs are observed afterwards. The subjects are divided according to age, gender, care with or without patch. In addition, a comparison with a control group that does not show any chronic or acute lung disease is made according to age and gender of the test group. In addition, in cooperation with the Division of Pediatric Pulmonology and Allergology of the Department of Pediatrics and Adolescent Medicine at the Medical University of Graz, the lung function of former diaphragmatic hernias patients (before administration of probiotics) and a control group is to be measured. In cooperation with the Medical Center of Sports Medicine the investigator also carry out a sports medical examination including ergospirometry. The duration of the study is set at 12 months.

Study participants: Study group: Children between 6-16 years of age, who are enrolled at the Department of Pediatric and Adolescent Surgery at the Medical University of Graz between 2000 and 2010 due to a congenital diaphragmatic hernia have received an operative closure with or without patch. Control group: Children between 6-16 years who do not have pulmonary disease. Recruited from the outpatient area at the Department of Pediatric and Adolescent Surgery at the Medical University of Graz. The aim is to establish contact with the above-mentioned patients and their parents and to achieve willingness to participate in this study by means of an information letter. The control group should come from the area of outpatient area in the Department of Pediatric and Adolescent Surgery, Medical University of Graz, after appropriate information and possible consent.

Microbiome analysis before treatment with a probiotic: Collection of sample material - in this case sputum - from the deep respiratory tract by induced sputum after inhalation of hypersaline saline solution with resulting provocation of cough. The sample is then deep-frozen. The Microbiome measurement is performed as a comparative 16S rDNA-based profile via chip-based next-generation sequencing as already published, analyzed using SnowMAn, Qiime and MOTHUR as well as the own "R"-based software. A sequencing depth of 5,000-10,000 reads per sample.

VOCs analysis before treatment with a probiotic: I) Taking of the exhaled gas samples: One sample from inspiration and two from expiration is taken from each subject (n = 3). For sampling investigator use an automatic sampling system that is directly connected to a capnometer. This system contains a so-called needle-trap microextraction (NTME) as a microextraction technique and meets the requirements of an optimal sampling on currently technically highest level. The exhaled gas samples obtained in this way are then sent to our cooperation partner, to the Institute for Breathing Gas Analysis at the University of Rostock for analysis. II) Analysis of exhaled gas samples: There, the exhaled gas samples are thermally transferred into the inert carrier gas stream (He) in an injector of a chromatograph. The substances are assigned according to their retention time in the chromatogram and their mass spectrum. Unknown Compounds in the exhaled gas are identified by comparison with a reference database based on the mass spectrum. Vital and laboratory data, as well as microbiological information, are taken from the patients' findings. III) Identification of biomarkers of exhaled gas samples: From the results of the patient measurements, those substances and substance concentrations are determined which are specific for study group 1 and group 2, i.e. compounds which are not present in the comparison group or only in significantly lower or higher concentrations. The selected volatile markers, as well as any volatile contaminants that may have been detected in the environment, are stored in an analytical reference database and, after elimination of the contamination, bundled into possibly disease-specific marker profiles. IV) Analysis of fecal samples: The fecal samples are also sent to the Institute for Breathing Gas Analysis of the University of Rostock for analysis and analyzed there after appropriate preconcentration by solid phase microextraction (SPME). V) Identification of biomarkers of fecal samples: This is done in analogy to the exhaled gas samples.

Lung function measurement before treatment with a probiotic: Measurement of lung function using spirometry and body plethysmography (Fa Jäger spirometer and body plethysmograph) and nitrogen washout process (N2-multiple breath washout, System Exhalyzer D and Spiroware 3.1, Eco Medics AG, Duernten, Switzerland). Spirometry and body plethysmography are performed according to published ERS/ATS Standards. The "multiple breath washout" method is performed under resting breathing and detects the Ventilation (in)homogeneity at the level of the functional residual capacity (= FRC = that lung volume that is still in the lungs after a calm spontaneous exhalation is left behind). The system consists of a flow meter, a fast analyzing gas measuring system, a gas administration system and the corresponding Computer analysis software. As a "foreign gas" it will be use 78% of the gas in air occurring nitrogen (N2). A flow-volume measurement is performed via an Ultrasonic flowmeter performed directly in the inhalation and exhalation flow of the test person/patient and via a laser O2 sensor using the side current measurement method and an infrared CO2 sensor in the main current measuring procedure (= directly in the patient's respiratory flow) the respective gas concentration. The N2 component is then indirectly measured via the O2 and CO2 concentration (N2 = 1 - O2 - CO2). During calm spontaneous breathing, the Patient on a snorkel mouthpiece via a bacterial filter through the flowmeter 100% oxygen and thus "washes" N2 out ("N2-multiple breath washout"). In doing so, the flow-volume curve of spontaneous breathing "online" is displayed on the screen and the measurement at Reaching a 1/40 (= 2.5%) of the initial nitrogen concentration is completed. After that, wait the subject is safe in the length of twice the duration of the measurement around the oxygen of exhaling. This is followed by the next measurement. A total of 3 measurements whose mean value serves as a result. The so-called "lung clearance index", which indicates the number of functional residual capacity lung volumes, which can be used to reduce the initial nitrogen concentration to a 1/40 after oxygenation was required. (LCI = quotient between exhaled volume and FRC). It expresses how long it takes for the inhaled gas (in our case the physiologically occurring nitrogen in the air) through inhalation of 100% oxygen. For healthy persons, this value is on average 7 and is significantly higher in lung patients. Further measuring parameters, which makes a statement about the peripheral airways proximal to the terminal bronchioles on the one hand and via the more distal azine airways on the other hand are calculated.

Sports medical examination: To exclude contraindications for ergometry, a 12-channel resting ECG and a resting blood pressure measurement (CombynTM Function & Spaces ECG, Academic Technologies) are performed at the beginning of the examination. After the anthropometric data (height, weight, BMI) have been collected, the muscle mass and fat mass are determined by multi-frequency impedance measurement in six body segments (CombynTM Function & Spaces ECG, Academic Technologies). The lung function is measured by means of small spirometry at rest and after exercise (Spirometer Oxycon Pro, Reiner). In order to determine cardiopulmonary performance, ergospirometry is performed on a bicycle (Excalibur Sport ergometer, Lode company; Oxycon Pro spiroergometry unit, Reiner company) with a gradual increase in stress up to subjective exhaustion. The evaluation of these data allows conclusions to be drawn about the performance-limiting system (cardiovascular system, lungs, musculature) in addition to the determination of aerobic performance.

Microbiome/VOCs analysis after treatment with a probiotic: After sampling for microbiome and VOC analysis and carrying out lung function measurements and sports medical examination, the participants in the study group will take a probiotic (Omnibiotic 6, purchased from the Allergosan Institute, dietary supplement) for a period of 3 months. Immediately afterwards and another month later, measurements of the pulmonary microbiome and the VOCs in the breath are taken.

ELIGIBILITY:
Inclusion Criteria:

* Age from 6-16 years
* Age 0-6 months at time of CDH-OP (except control group)
* reliable diagnosis of congenital diaphragmatic hernia (except control group)
* surgical occlusion with patch (except control group)
* surgical occlusion without patch (except control group)
* given approval

Exclusion Criteria:

* chronic pulmonary diseases
* Infection within 4 weeks before the test date
* unaccepted consent

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Analysis of the pulmonary microbiome in the sputum of CDH group versus control group. | 12 months
  OTUs (Operational Taxonomic Units) will be visualized as OTU tables, bar charts and PCOA (Principal Coordinates Analysis) plots using the Qiime core microbiome script. For the different groups alpha-diversity (Chao 1 index, Shannon Index etc.) will be compared. Additionally, we will compare beta-diversity by Adonis test. Relative abundances of the bacteria at the different levels (phylum to genus) will be compared between the groups by using Kruskal Wallis Test.
Analysis of VOCs in the respiratory air by needle-trap microextraction (NTME) and stool by solid phase microextraction (SPME) of CDH group versus control group. | 12 months
  From the results of the patient measurements, those substances and substance concentrations are determined which are specific for study group 1 and group 2, i.e. compounds which are not present in the comparison group or only in significantly lower or higher concentrations. The selected volatile markers, as well as any volatile contaminants that may have been detected in the environment, are stored in an analytical reference database and, after elimination of the contamination, bundled into possibly disease-specific marker profiles. The VOCs are recorded and displayed in the following order. The unit in which the VOCs are measured is pars per billion (ppb).
  Class (for example carbons) VOCs (ppb) CDHV1 (congenital diaphragmatic hernia group visit 1) CDHK (congenital diaphragmatic hernia - control group visit 1) CDHV2 (congenital diaphragmatic hernia group visit 2) CDHV3 (congenital diaphragmatic hernia group visit 3) p-value
Analysis of the lung function: Lung clearance index (LCI) is derived from multiple breath washout tests of CDH group versus control group. | 12 months
  The LCI is about 7 (range from 6.45-7.78) for healthy individuals and is a number without a unit.
Analysis of the lung function: Forced expiratory volume in one second (FEV1) measured with spirometry of CDH group versus control group. | 12 months
  The FEV1 is the forced expiratory volume within the first second (liter/second), generated by a maximal voluntary exhalation after maximum inspiration before, usually described as the Tiffeneau-Index in % of FVC (FEV1/FVC).
Analysis of the cardiopulmonary capacity: Resting ECG of CDH group versus control group. | 12 months
  A Resting ECG recording the resting heart rate, the rhythm, the PQ duration, the width and height of the QRS complex, the QT duration, and the ST segment is recorded.
Analysis of the cardiopulmonary capacity: Systolic and diastolic blood pressures of CDH group versus control group. | 12 months
  Noninvasiv systolic and diastolic blood pressures are assessed (Unit: mmHg).
Analysis of the cardiopulmonary capacity: Body height of CDH group versus control group. | 12 months
  Body height is measured in cm.
Analysis of the cardiopulmonary capacity: Body weight of CDH group versus control group. | 12 months
  Body weight is measured in kg.
Analysis of the cardiopulmonary capacity: Body mass index (BMI) of CDH group versus control group. | 12 months
  Body mass index is calculated in kg body weight/body height².
Analysis of the cardiopulmonary capacity: Muscle mass of CDH group versus control group. | 12 months
  Muscle mass is specified in kg/body height².
Analysis of the cardiopulmonary capacity: Body fat of CDH group versus control group. | 12 months
  Body fat is specified in percent of body weight.
Analysis of the cardiopulmonary capacity: Aerobic performance of CDH group versus control group. | 12 months
  Aerobic performance is specified in percent of normal values of the Austrian cardiological society.
Analysis of the cardiopulmonary capacity: Maximal oxygen uptake of CDH group versus control group. | 12 months
  Measurements by spiroergometry: Maximal oxygen uptake in ml/kg/min.
Analysis of the cardiopulmonary capacity: Ventilation of CDH group versus control group. | 12 months
  Measurements by spiroergometry: Ventilation in liter/min.
Analysis of the cardiopulmonary capacity: Oxygen pulse of CDH group versus control group. | 12 months
  Measurements by spiroergometry: Oxygen pulse in ml/beats per minute.
Analysis of the cardiopulmonary capacity: Oxygen uptake of CDH group versus control group. | 12 months
  Respiratory exchange ratio = oxygen uptake in ml/carbon dioxide release in ml.
Analysis of the cardiopulmonary capacity: Breathing reserve of CDH group versus control group. | 12 months
  Unit: Percent of FEV1 x 35.

SECONDARY OUTCOMES:
Alterations of pulmonary microbiome after probiotic treatment for a period of 3 months in patients with CDH. | 12 months
  After sampling for microbiome and VOC analysis and carrying out lung function measurements and sports medical examination, the participants in the study group will take a probiotic (Omnibiotic 6, purchased from the Allergosan Institute, dietary supplement) for a period of 3 months. Immediately afterwards and another month later, measurements of the pulmonary microbiome are taken.
Alterations of VOCs in the respiratory air after probiotic treatment for a period of 3 months in patients with CDH. | 12 months
  After sampling for microbiome and VOC analysis and carrying out lung function measurements and sports medical examination, the participants in the study group will take a probiotic (Omnibiotic 6, purchased from the Allergosan Institute, dietary supplement) for a period of 3 months. Immediately afterwards and another month later, measurements of the VOCs in the breath are taken.
Analysis of the lung function: Forced expiratory flow (FEF25-75). | 12 months
  Measured by body plethysmography and spirometry: FEF25-75 = Forced expiratory flow 25-75% vital capacity (= MMEF), Unit: l/s.
Analysis of the lung function: Forced expiratory flow (FEF25). | 12 months
  Measured by body plethysmography and spirometry: FEF25 = Forced expiratory flow at the time, when 75% of the vital capacity is exhaled (MEF25), Unit: l/s.
Analysis of the lung function: Forced expiratory flow (FEF50). | 12 months
  Measured by body plethysmography and spirometry: FEF50 = Forced expiratory flow at 50% of the exhaled vital capacity (= MEF50), Unit: l/s.
Analysis of the lung function: Forced expiratory volume (FEV1). | 12 months
  Measured by body plethysmography and spirometry: FEV1 = Forced expiratory volume in 1 s, Unit: l.
Analysis of the lung function: Tiffeneau-Index (FEV1%FVC). | 12 months
  Measured by body plethysmography and spirometry: FEV1%FVC = Tiffeneau-Index, described in % of the forced vital capacity, Unit: %.
Analysis of the lung function: Functional residual capacity (FRC). | 12 months
  Measured by body plethysmography and spirometry: FRC = Functional residual capacity, Unit: l.
Analysis of the lung function: Through "multiple breath washout" acquired FRC (RC(MBW)). | 12 months
  RC(MBW): Through "multiple breath washout" acquired FRC, Unit: l.
Analysis of the lung function: Through body plethysmography acquired FRC (RC(pleth)). | 12 months
  Measured by body plethysmography: RC(pleth): Through body plethysmography acquired FRC (= ITGV, intra thoracic gas volume), Unit: l.
Analysis of the lung function: Forced vital capacity (FVC). | 12 months
  Measured by spirometry: FVC = Forced vital capacity, Vital capacity acquired through a forced exhaled manoeuvre, Unit: l.
Analysis of the lung function: Intrathoracic gasvolume (ITGV). | 12 months
  Measured by body plethysmography: ITGV = Intrathoracic gasvolume (= FRC(pleth)), Unit: l.
Analysis of the lung function: Max. expiratory flow (MEF25). | 12 months
  Measured by spirometry: MEF25 = Max. expiratory flow when 75% of the vital capacity is exhaled (= FEF25), Unit: l/s.
Analysis of the lung function: Max. expiratory flow (MEF50). | 12 months
  Measured by spirometry: MEF50 = Max. expiratory flow when 50% of the vital capacity is exhaled (= FEF50), Unit: l/s.
Analysis of the lung function: Max. expiratory flow (MMEF). | 12 months
  Measured by spirometry: MMEF = Max. expiratory flow (= FEF25-75), Unit: l/s.

CONTACTS AND LOCATIONS:
Overall Officials: Till Holger, MD, Study Director — Department of Pediatric and Adolescent Surgery, Medical University of Graz; Ernst Eber, MD, Principal Investigator — Department of Pediatric and Adolescent Medicine, Medical University of Graz; Gert Warncke, MD, Principal Investigator — Department of Pediatric and Adolescent Surgery, Medical University of Graz
Locations (1):
- Department of Department of Pediatric and Adolescent Surgery, Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kotecha S, Barbato A, Bush A, Claus F, Davenport M, Delacourt C, Deprest J, Eber E, Frenckner B, Greenough A, Nicholson AG, Anton-Pacheco JL, Midulla F. Congenital diaphragmatic hernia. Eur Respir J. 2012 Apr;39(4):820-9. doi: 10.1183/09031936.00066511. Epub 2011 Oct 27. PMID 22034651
- [Background] Tracy M, Cogen J, Hoffman LR. The pediatric microbiome and the lung. Curr Opin Pediatr. 2015 Jun;27(3):348-55. doi: 10.1097/MOP.0000000000000212. PMID 25888147
- [Background] Caverly LJ, Zhao J, LiPuma JJ. Cystic fibrosis lung microbiome: opportunities to reconsider management of airway infection. Pediatr Pulmonol. 2015 Oct;50 Suppl 40:S31-8. doi: 10.1002/ppul.23243. PMID 26335953
- [Background] Bergmann A, Trefz P, Fischer S, Klepik K, Walter G, Steffens M, Ziller M, Schubert JK, Reinhold P, Kohler H, Miekisch W. In Vivo Volatile Organic Compound Signatures of Mycobacterium avium subsp. paratuberculosis. PLoS One. 2015 Apr 27;10(4):e0123980. doi: 10.1371/journal.pone.0123980. eCollection 2015. PMID 25915653
- [Background] Fischer S, Trefz P, Bergmann A, Steffens M, Ziller M, Miekisch W, Schubert JS, Kohler H, Reinhold P. Physiological variability in volatile organic compounds (VOCs) in exhaled breath and released from faeces due to nutrition and somatic growth in a standardized caprine animal model. J Breath Res. 2015 May 14;9(2):027108. doi: 10.1088/1752-7155/9/2/027108. PMID 25971714
- [Background] Pereira J, Porto-Figueira P, Cavaco C, Taunk K, Rapole S, Dhakne R, Nagarajaram H, Camara JS. Breath analysis as a potential and non-invasive frontier in disease diagnosis: an overview. Metabolites. 2015 Jan 9;5(1):3-55. doi: 10.3390/metabo5010003. PMID 25584743
- [Background] Amann A, Costello Bde L, Miekisch W, Schubert J, Buszewski B, Pleil J, Ratcliffe N, Risby T. The human volatilome: volatile organic compounds (VOCs) in exhaled breath, skin emanations, urine, feces and saliva. J Breath Res. 2014 Sep;8(3):034001. doi: 10.1088/1752-7155/8/3/034001. Epub 2014 Jun 19. PMID 24946087
- [Background] Barker M, Hengst M, Schmid J, Buers HJ, Mittermaier B, Klemp D, Koppmann R. Volatile organic compounds in the exhaled breath of young patients with cystic fibrosis. Eur Respir J. 2006 May;27(5):929-36. doi: 10.1183/09031936.06.00085105. Epub 2006 Feb 2. PMID 16455833
- [Background] Miekisch W, Schubert JK, Noeldge-Schomburg GF. Diagnostic potential of breath analysis--focus on volatile organic compounds. Clin Chim Acta. 2004 Sep;347(1-2):25-39. doi: 10.1016/j.cccn.2004.04.023. PMID 15313139
- [Background] Forton J. Induced sputum in young healthy children with cystic fibrosis. Paediatr Respir Rev. 2015 Oct;16 Suppl 1:6-8. doi: 10.1016/j.prrv.2015.07.007. Epub 2015 Sep 26. PMID 26410282
- [Background] Planting NS, Visser GL, Nicol MP, Workman L, Isaacs W, Zar HJ. Safety and efficacy of induced sputum in young children hospitalised with suspected pulmonary tuberculosis. Int J Tuberc Lung Dis. 2014 Jan;18(1):8-12. doi: 10.5588/ijtld.13.0132. PMID 24365546
- [Background] Marri PR, Stern DA, Wright AL, Billheimer D, Martinez FD. Asthma-associated differences in microbial composition of induced sputum. J Allergy Clin Immunol. 2013 Feb;131(2):346-52.e1-3. doi: 10.1016/j.jaci.2012.11.013. Epub 2012 Dec 23. PMID 23265859
- [Background] Gorkiewicz G, Thallinger GG, Trajanoski S, Lackner S, Stocker G, Hinterleitner T, Gully C, Hogenauer C. Alterations in the colonic microbiota in response to osmotic diarrhea. PLoS One. 2013;8(2):e55817. doi: 10.1371/journal.pone.0055817. Epub 2013 Feb 8. PMID 23409050
- [Background] Trefz P, Rosner L, Hein D, Schubert JK, Miekisch W. Evaluation of needle trap micro-extraction and automatic alveolar sampling for point-of-care breath analysis. Anal Bioanal Chem. 2013 Apr;405(10):3105-15. doi: 10.1007/s00216-013-6781-9. Epub 2013 Feb 7. PMID 23388692
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Wanger J, Clausen JL, Coates A, Pedersen OF, Brusasco V, Burgos F, Casaburi R, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson D, Macintyre N, McKay R, Miller MR, Navajas D, Pellegrino R, Viegi G. Standardisation of the measurement of lung volumes. Eur Respir J. 2005 Sep;26(3):511-22. doi: 10.1183/09031936.05.00035005. No abstract available. PMID 16135736